CLINICAL TRIAL: NCT05235165
Title: A Phase 3 Randomized Controlled Trial Comparing Open vs Thoracoscopic Management of Pulmonary Metastases in Patients With Osteosarcoma
Brief Title: Thoracotomy Versus Thoracoscopic Management of Pulmonary Metastases in Patients With Osteosarcoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOST2031; NCI-2021-14237 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AOST2031 (Other: Children's Oncology Group); AOST2031 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2022-01-19; First posted 2022-02-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Malignant Neoplasm in the Lung; Metastatic Osteosarcoma; Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Specimen Handling; Thoracoscopy; Thoracotomy; Thoracostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm A (thoracotomy) (Experimental): Patients undergo open thoracic surgery (thoracotomy). Patients undergo CT throughout the trial. Patients may also undergo collection of tissue on study and blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Questionnaire Administration; Procedure: Thoracotomy
- Arm B (thoracoscopy) (Experimental): Patients undergo thoracoscopy (video-assisted thoracoscopic surgery or VATS). Patients undergo CT throughout the trial. Patients may also undergo collection of tissue on study and blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration; Procedure: Thoracoscopy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue and blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
  Arms: Arm A (thoracotomy)
Other: Questionnaire Administration — Ancillary studies
Procedure: Thoracoscopy — Undergo video-assisted thoracoscopic surgery or VATS
  Other Names: Pleuroscopy
  Arms: Arm B (thoracoscopy)
Procedure: Thoracotomy — Undergo open thoracic surgery
  Other Names: incision of Chest Wall; Incision of Thorax
  Arms: Arm A (thoracotomy)

SUMMARY:
This phase III trial compares the effect of open thoracic surgery (thoracotomy) to thoracoscopic surgery (video-assisted thoracoscopic surgery or VATS) in treating patients with osteosarcoma that has spread to the lung (pulmonary metastases). Open thoracic surgery is a type of surgery done through a single larger incision (like a large cut) that goes between the ribs, opens up the chest, and removes the cancer. Thoracoscopy is a type of chest surgery where the doctor makes several small incisions and uses a small camera to help with removing the cancer. This trial is being done evaluate the two different surgery methods for patients with osteosarcoma that has spread to the lung to find out which is better.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if open surgical resection is superior to thoracoscopic resection for thoracic event-free survival (tEFS) in patients with resectable oligometastatic pulmonary osteosarcoma.

SECONDARY OBJECTIVES:

I. To determine if open surgical resection is superior to thoracoscopy for event free survival (EFS) in patients with resectable oligometastatic pulmonary osteosarcoma.

II. To determine if open surgical resection is superior to thoracoscopy for overall survival (OS) in patients with resectable oligometastatic pulmonary osteosarcoma.

III. To determine if thoracoscopy is superior to open surgical resection for post-operative pain interference in patients with resectable oligometastatic pulmonary osteosarcoma.

EXPLORATORY OBJECTIVES:

I. To compare 30-day rates of perioperative surgical complications for both open surgical resection and thoracoscopy.

II. To compare patterns of recurrence (ipsilateral and/or contralateral) in patients who undergo open or thoracoscopic resection for unilateral or bilateral pulmonary metastases.

III. To describe the use of localization techniques and its relationship with both surgical approach and pathologic findings.

IV. To assess the prognostic significance of a decision to change the post-operative treatment plan.

V. To describe the relationship between the preoperative chest computed tomography (CT) imaging, intraoperative surgical findings, and pathologic results, comparing radiological features to the presence of viable tumor.

VI. To prospectively compare between treatment arms the relationship between surgical approach and patient-reported outcomes (PROs), specifically patient functional impairment of the upper extremities, pain intensity, and health-related quality of life (HRQoL).

VII. To generate well-characterized, clinically-annotated, distributable models of metastatic osteosarcoma.

VIII. To collect and bank pulmonary metastatic lesions (including frozen tissues and paired metastatic lesions coming from the same patient) to facilitate study of metastatic disease and serial blood samples for future tumor profiling, germline and circulating tumor deoxyribonucleic acid (DNA) studies.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM A: Patients undergo open thoracic surgery (thoracotomy).

ARM B: Patients undergo thoracoscopy (video-assisted thoracoscopic surgery or VATS).

All patients undergo computed tomography (CT) throughout the trial. Patients may also undergo collection of tissue on study and blood throughout the trial.

After completion of study treatment, patients are followed up at 7-14 days, 4-6 weeks, and 3 months post-surgery and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be < 50 years at the time of enrollment.
* Patients must have =< 4 nodules per lung consistent with or suspicious for metastases, with at least one of which being >= 3 mm and all of which must be =< 3 cm size.

  * Note: Patient must have eligibility confirmed by rapid central imaging review.
* Lung nodules must be considered resectable by either open thoracotomy or thoracoscopic surgery. Determination of resectability is made by the institutional surgeon.
* Patients must have a histological diagnosis of osteosarcoma.
* Patients must have evidence of metastatic lung disease at the time of initial diagnosis, or at time of 1st recurrence following completion of therapy for initially localized disease.
* Patients with newly diagnosed disease must have completed successful gross tumor resection for their primary tumor or surgical local control of primary tumor must be planned to be performed simultaneously with thoracic surgery.
* Newly diagnosed patients must be receiving or recently completed (within 60 days) systemic therapy considered by the treating physician to be standard treatment for newly diagnosed osteosarcoma (eg, cisplatin-doxorubicin or ifosfamide-based drug regimens) at the time of enrollment on this study. Dose and drug modifications for toxicity do not exclude patients from participation.
* Patients at time of 1st recurrence must have completed systemic therapy for their initial primary tumor, considered by the treating physician to be standard treatment for newly diagnosed osteosarcoma (eg, cisplatin-doxorubicin or ifosfamide-based drug regimens) at the time of enrollment on this study. Dose and drug modifications for toxicity do not exclude patients from participation.

Exclusion Criteria:

* Patients with unresectable primary tumor.
* Patients with pulmonary metastatic lesions that would require anatomic resection (lobectomy or pneumonectomy) or lesions that are defined as "central" (i.e., central lesion involves or is proximal to segmental bronchi and peripheral is lesion distal to segmental bronchi).
* Patients with chest wall or mediastinal based metastatic lesions, or with significant pleural effusion.
* Patients with disease progression at either the primary or pulmonary metastatic site while on initial therapy. Note: Once the patient has been enrolled on the study, additional computed tomography (CT) scans are not anticipated prior to thoracic surgery. Note: Some variation in nodule size measurements over the course of pre-operative therapy is anticipated and does not qualify for exclusion unless deemed true disease progression by the primary treatment team.
* Patients with evidence of extrapulmonary metastatic disease.
* Patients who received therapeutic pulmonary surgery for lung metastasis prior to enrollment.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Thoracic event-free survival (tEFS) | Four years after enrollment
  Estimated four year thoracic event free survival (tEFS) where tEFS is calculated as the time from study enrollment. Any recurrence within the pulmonary parenchyma, involving the pleural surface or the drain/surgical site wound will be considered an event. A death that results from the procedure, as confirmed by the treating physician, will be considered an event. Patients with recurrences arising outside the thoracic region, the diagnosis of a malignancy that is not osteosarcoma (SMN) or death considered unrelated to the study surgical procedure, as confirmed by the treating physician will be considered competing events provided these occur prior to a thoracic cavity event as defined above. Patients without an event of any kind at last contact are considered censored.

SECONDARY OUTCOMES:
Event free survival (EFS) | Four years after enrollment
  Estimated four year EFS where EFS is calculated as the time from study enrollment to disease progression, disease relapse, occurrence of a second malignant neoplasm, death from any cause or last follow-up whichever occurs first. Patients without an event at last contact are considered censored.
Overall survival (OS) | Four years after enrollment
  Time from study enrollment to death or last patient contact. Patients alive at last contact are considered censored.
Post operative pain interference at time point 3, 7-14 days after surgical intervention | 7-14 days after surgical intervention
  Total PROMIS pain interference score from the 8 item PROMIS pain interference short form.
Post operative pain interference at time point 4, 4-6 weeks after surgical intervention | 4-6 weeks after surgical intervention
  Total PROMIS pain interference score from the 8 item PROMIS pain interference short form.

OTHER OUTCOMES:
Perioperative surgical complications | At 30 days post-op
  The descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 will be utilized for AE reporting.
Mode of tEFS event | Four years after enrollment
  Classified as: (1) ipsilateral recurrence site; (2) contralateral recurrence site; or (3) ipsilateral and contralateral recurrence site. The analysis will be restricted to patients with unilateral disease at enrollment.
Use of localization techniques | 12 months after enrollment
  Data collection will include a description of all localization methods used.
Decision to change the post-operative treatment plan | 12 months after enrollment
  Whether the investigator adhered to the post-thoracic surgery plan for systemic therapy.
Radiological features to the presence of viable tumor | 12 months after enrollment
  Radiological features and pathological characteristics of lung nodules contributed by the same patient.
Post operative upper extremity function at time point 2, 24-48 hours after surgical intervention | 24-48 hours after surgical intervention
  Total PROMIS upper extremity score from the 8 item PROMIS upper extremity short form.
Post operative upper extremity function at time point 3, 7-14 days after surgical intervention | 7-14 days after surgical intervention
  Total PROMIS upper extremity score from the 8 item PROMIS upper extremity short form.
Post operative pain intensity at time point 2, 24-48 hours after surgical intervention | 24-48 hours after surgical intervention
  NRS 11 single item pain intensity score.
Post operative pain intensity at time point 3, 7-14 days after surgical intervention | 7-14 days after surgical intervention
  NRS 11 single item pain intensity score.
Frequency of obtaining quality tumor tissue for biological analysis | 1 month after surgical intervention
  Tumor samples obtained from the surgical procedure that are submitted to the COG tissue bank and subjected to dual nucleic acid extraction will be classified by central review as to whether sufficient tumor content was obtained for ultra low passage whole genome sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: John J Doski, Principal Investigator — Children's Oncology Group
Locations (232):
- United States (219):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Northern Nevada Radiation Oncology, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Westchester Medical Center, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Valley Medical Center, Renton, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia